CLINICAL TRIAL: NCT03028155
Title: Concentration-based Versus Body Surface Area-based Peroperative Intraperitoneal Chemotherapy (HIPEC) After Optimal Cytoreductive Surgery in Colorectal Peritoneal Carcinomatosis' Treatment - Randomized Non-blinded Phase III Clinical Trial
Brief Title: Concentration- Versus Body Surface Area-based HIPEC in Colorectal Peritoneal Carcinomatosis' Treatment
Acronym: COBOX
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hasselt University (Other)
Collaborators: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Principal Investigator, Kurt Van der Speeten, prof. dr., Hasselt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZOLCOBOX1
Record Dates: First submitted 2016-12-24; First posted 2017-01-23 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Colorectal Peritoneal Carcinomatosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxaliplatin: BSA-based HIPEC (Active Comparator): Intervention: oxaliplatin: BSA-based HIPEC HIPEC will be performed using oxaliplatin as chemotherapeutic agent at a dose of 460 mg/m2 mixed in 0.9% saline carrier solution during 30 minutes. Volume of the carrier solution: depended on the capacity of the abdominal cavity of the patient.
  Interventions: Drug: Oxaliplatin: BSA-based HIPEC
- Oxaliplatin: Concentration-based HIPEC (Active Comparator): Intervention: oxaliplatin: concentration-based HIPEC HIPEC will be performed using oxaliplatin as chemotherapeutic agent at a dose of 460 mg/m2 mixed in 0.9% saline carrier solution at 2L/m2, which equals a concentration of 230 mg/L during 30 minutes.
  Interventions: Drug: Oxaliplatin: Concentration-based HIPEC

INTERVENTIONS:
Drug: Oxaliplatin: BSA-based HIPEC — oxaliplatin: 460 mg/m2 volume: dependent on the capacity of the peritoneal cavity of the patient
  Arms: Oxaliplatin: BSA-based HIPEC
Drug: Oxaliplatin: Concentration-based HIPEC — oxaliplatin: 230 mg/L
  Arms: Oxaliplatin: Concentration-based HIPEC

SUMMARY:
Colorectal Cancer (CRC) is the third most common cancer and the fourth most common cause of cancer-related death worldwide. CRC frequently gives rise to transcoelomic spread of tumor cells in the peritoneal cavity, which ultimately leads to Peritoneal Carcinomatosis (PC). A new loco-regional treatment modality combines Cytoreductive Surgery (CRS) and Hyperthermic Intraperitoneal Peroperative Chemotherapy (HIPEC). The current HIPEC dosing regimens for the treatment of colorectal PC can be divided into body surface area (BSA)-based protocols and concentration-based protocols. Most groups currently use a drug dose based on calculated BSA (mg/m2) in analogy to systemic chemotherapy regimens. These regimens take BSA as a measure for the effective contact area, represented as the peritoneal surface in the formula for dose intensification. However, an imperfect correlation exists between actual peritoneal surface area and calculated BSA. Sex differences, but also altered pathophysiological characteristics or frequent complications in patients (ascites) are responsible for differences in peritoneal surface areas, which in turn affect absorption characteristics. This takes us away from the initial homogenous drug concentration desired, increasing the variability in the systemic and tumor exposure to the drug. Pharmacokinetic changes induced by the volume of chemotherapy solution with constant drug dose, administered intraperitoneally, have already been reported. This resulted in less precise predictions of the toxicity associated with the treatment. By contrast, some groups use a totally different dosimetry regimen based on concentration. From a pharmacologic point of view, the big advantage of a concentration-based system is that the residual tumor nodules after CRS are exposed to a constant diffusional force and, thus, cytotoxicity. Unfortunately the prize to be paid for a better prediction of the efficacy of the IP chemotherapy is a high unpredictability of the levels of plasmatic cancer chemotherapy and, thus, toxicity. This randomised non-blinded phase III clinical trial will be the first trial to pharmacologically evaluate the two dosing regimens, BSA-based and concentration-based, both applied as standard of care in current practice.

ELIGIBILITY:
Inclusion Criteria:

* Males and females with histologically proven synchronous or metachronous peritoneal metastases from colorectal origin
* Karnofsky index > 70%
* Age >18 years
* Fit for major surgery
* Mentally capable of understanding the proposed treatment and the provided informed consent
* Estimated life expectancy of > 6 months
* Absence of other malignant disease
* Serum creatinine < or = 1.5 mg/dL or calculated glomerular filtration rate > or = 60 mL/min/1.73m2
* Serum total bilirubin < or = 1.5 mg/dL except for known Gilbert's disease
* Platelet count > 100,000/µL
* Hemoglobin > 9 g/dL
* Neutrophil granulocytes > 1,500/mL
* International normalized ratio < or = 2

Exclusion Criteria:

* Alcohol or drug abuse
* Inclusion in other trials interfering with the study protocol
* Chronic systemic immune therapy
* Chemotherapy or hormone therapy not indicated in the study protocol
* Severe organ insufficiency
* Pregnancy or breast feeding
* Appearance of distant metastases (liver, lung) of a CT scan of the abdomen of chest X-ray
* Severe or uncontrolled cardiac pathology
* > 6 months occurrence of myocardial infarction
* Presence of congestive cardiac failure of symptomatic angor pectoris despite optimal medical treatment
* Presence of congestive cardiac failure of cardiac arrhythmia requiring medical treatment with insufficient rhythm control
* Uncontrolled arterial hypertension
* Active bacterial, viral or fungal infection
* Active gastrointestinal ulcer
* Any stage cirrhosis
* Uncontrolled diabetes mellitus
* Severe obstructive or restrictive respiratory insufficiency
* Tumor in the presence of obstruction
* Allergy to trial related drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Assessment of pharmacologic advantage | Day 2
  the area-under-the-curve (AUC) ratio of the intraperitoneal (IP) exposure over the AUC of the intravenous (IV) exposure to oxaliplatin. Intraoperative sampling of plasma and peritoneal fluid at seven time points (0, 5, 10, 15, 20, 25 and 30 minutes) during the 30-minute HIPEC procedure.
  The concentration of oxaliplatin will be determined in plasma and peritoneal fluid by means of a validated inductively coupled plasma mass spectrometry (ICP-MS). A concentration versus time curve will be set-up and the AUC will be determined.
Assessment of Pt excretion in urine | day 2
  Intraoperative sampling of urine at seven time points (0, 5, 10, 15, 20, 25 and 30 minutes) during the 30-minute HIPEC procedure. The concentration of oxaliplatin will be determined in urine by means of a validated ICP-MS. A concentration versus time curve will be set-up and the AUC will be determined.
Assessment of efficacy in the tumor nodule as pharmacologic endpoint. | day 2
  At the day of surgery (day 2): intraoperative sampling of tumor nodules at seven time points (0, 5, 10, 15, 20, 25 and 30 minutes) during the 30-minute HIPEC procedure. The concentration of oxaliplatin will be determined in tumor nodules by means of a validated ICP-MS. A concentration versus time curve will be set-up and the AUC will be determined.
Assessment of 3-month overall morbidity and mortality | During 3 months postoperative.
  Morbidity and mortality will be evaluated using the Clavien-Dindo classification. This classification consists of five grades: grade I, deviation from standard post-operative course within 'allowed therapeutic regimens'; grade II, complication requiring surgical, endoscopic or radiological intervention; grade IV, complication requiring ICU admission and grade V, complication resulting in death.

SECONDARY OUTCOMES:
Assessment of one-year overall survival | During one year postoperative.
  One-year overall survival will be determined.
Assessment of health related quality of life (HRQOL): EORTC QLQ-C-30 | Day 1
  HRQOL will be determined by means of the EORTC QLQ-C-30 (version 3.0, 2001). This questionnaire is developed to evaluate quality of life (QOL) of cancer patients, translated and validated in Dutch. Scoring will be according to manufacturer's guidelines, EORTC scoring manual.
Assessment of health related quality of life (HRQOL): SF-36 | Day 1
  HRQOL will be determined by means of the 36-item Short Form Survey (SF-36). This questionnaire is developed by RAND Health. Scoring will be according to instructions form RAND Health.
Assessment of health related quality of life (HRQOL): EORTC QLQ-C-30 | up to 2 months
  HRQOL will be determined by means of the EORTC QLQ-C-30 (version 3.0, 2001). This questionnaire is developed to evaluate quality of life (QOL) of cancer patients, translated and validated in Dutch. Scoring will be according to manufacturer's guidelines, EORTC scoring manual.
Assessment of health related quality of life (HRQOL): SF-36 | up to 2 months
  HRQOL will be determined by means of the 36-item Short Form Survey (SF-36). This questionnaire is developed by RAND Health. Scoring will be according to instructions form RAND Health.
Assessment of health related quality of life (HRQOL): EORTC QLQ-C-30 | month 3
  HRQOL will be determined by means of the EORTC QLQ-C-30 (version 3.0, 2001). This questionnaire is developed to evaluate quality of life (QOL) of cancer patients, translated and validated in Dutch. Scoring will be according to manufacturer's guidelines, EORTC scoring manual
Assessment of health related quality of life (HRQOL): SF-36 | month 3
  HRQOL will be determined by means of the 36-item Short Form Survey (SF-36). This questionnaire is developed by RAND Health. Scoring will be according to instructions form RAND Health.

CONTACTS AND LOCATIONS:
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Belgium

IPD SHARING:
Plan to Share IPD: No